CLINICAL TRIAL: NCT04038658
Title: Move-It: A Cluster-randomised Digital Worksite Exercise Intervention in China: Outcome and Process Evaluation
Brief Title: Digital Worksite Exercise Intervention in China: Outcome and Process Evaluation
Acronym: Move-It
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Holly Blake, Dr Holly Blake, Associate Professor, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Lai/27/6/13
Record Dates: First submitted 2019-07-23; First posted 2019-07-31 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Physical Activity
Keywords: exercise; worksite; digital; health promotion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster randomised control trial
Who Masked: Outcomes Assessor
Masking Description: Statistical analysis undertaken by researcher blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (MoveIt) (Experimental): 10-minute Qigong exercise session (video demonstration via website) delivered twice a day at set break times during the working day for 12 consecutive weeks
  Interventions: Behavioral: Move-It
- Wait-list control group (No Intervention): No intervention for 12 weeks. Then received the MoveIt Intervention for 12 weeks.

INTERVENTIONS:
Behavioral: Move-It
  Arms: Intervention Group (MoveIt)

SUMMARY:
The aim of the study is to evaluate the outcomes and processes of a video and web-based worksite exercise intervention for sedentary office workers in China.

The intervention is informed by behaviour change theory, and is a digital workplace intervention (called Move-It) involving a 10-minute Qigong exercise session (video demonstration via website) which is delivered twice a day at set break times during the working day for 12 consecutive weeks.

The setting is a large organisation with 2 sites (in Beijing and Guangzhou). The objectives are to examine the effect of a video-based intervention on employees' physical activity, time spent sitting and work performance. This is tested in a 2-group, randomised wait-list control trial. This means that employees at one site receive the intervention first (site 1 - intervention group), and when they have completed (12 weeks later), the other site then receives the same intervention (site 2 - wait-list control). At the end of the intervention, there is a process evaluation with the intervention group which includes focus groups with employees and managers to gather information about the way in which the intervention was implemented. The process evaluation is based on a framework called 'Reach Effectiveness Adoption Implementation Maintenance' (RE-AIM). Data were collected at baseline (before the intervention began) and after 12 weeks in both groups.

DETAILED DESCRIPTION:
Aim The aim of the study is to deliver a digital video-based worksite exercise intervention in China and conduct outcome and process evaluation. The objectives are: [1] to examine the effect of a video-based intervention on physical activity (PA) and weekday sitting hours (individual level); [2] to examine the effect of a video-based intervention on individual work performance (individual level); [3] to conduct a process evaluation of the intervention implementation (individual and cluster level).

Design This is a 2-arm cluster-randomised wait-list control trial, with outcomes assessed in two groups: intervention and wait-list control (objectives 1 and 2).

Clusters (sites) will be randomly allocated to groups at 1:1 ratio using computer-generated random number sequence.

Setting 2 sites of a major organisation in China (one in Beijing, one in Guangzhou), with a total of 490 employees.

Data Collection Data will be collected through online questionnaires emailed to all employee participants (Time 1 = T1). Employees in both groups will complete a second online questionnaire (Time 2 = T2). For the intervention group T2 will be immediately post-intervention, for the wait-list control group this will be just prior to receiving the intervention.

Sample size At an individual level, the estimated sample size is a minimum 72 for intervention group and 72 for control group, alpha 0.05, beta 0.2 and power 0.8.

Intervention This digital intervention consists of a series of six video clips demonstrating Qigong exercises designed to be undertaken at set exercise break times during the working day. The intervention includes a specially designed logo and selected images to be used on promotional posters and a dedicated 'Move-It' webpage. The six promotional videos are designed to be posted in sequence, one every two weeks, on the Move-It website. A Move-It icon on each employee's desktop computer screen will be scheduled to pop up twice a day as a prompt to interrupt sitting. The intervention is designed to be completed within 12 weeks.

Measures Self-report measures of PA, work performance and weekday sitting hours are taken at T1 (baseline) and T2 (12 week follow-up).

Data analysis Intervention outcome data will be analysed using the Statistical Package for the Social Sciences (IBM SPSS) Version 24.

Outcomes will be compared between the pre- and post-intervention time points. Intracluster correlations and estimated effects sizes will be presented for each outcome. Data from both clusters will be included in all analyses, and analysis is by intention-to-treat.

Process evaluation Will take place at the end of the intervention (intervention site only). This will include up to 6 focus groups (up to n=35) with employees (both participants and non-participants), organisational committee members and senior management.

These will be aligned with the RE-AIM framework to explore intervention reach, effectiveness, adoption, implementation and maintenance.

ELIGIBILITY:
Inclusion Criteria:

Employee of participating organisation

Exclusion Criteria:

Not an employee of participating organisation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2013-10-07 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) Taiwanese short form | Covers a person's record of physical activity for a period of seven days
  Measure of self-reported physical activity. Includes culturally sensitive Chinese translations for the terms "moderate", "vigorous" and "physical activity" as well as to identify representative types of physical activity for Taiwanese. Content validity 0.994.

SECONDARY OUTCOMES:
Health and Work Performance Questionnaire (HPQ). | Overall performance rating for the days worked over the past 4 weeks.
  Self-reported work performance. Single item was used from this scale. Item was measured on a 10-point scale ranging from 0=worst performance to 10=top performance.
  Item is: 'how would you rate your overall performance on the days you worked during the past 4 weeks?'.
Weekday sitting hours | 1 day (average)
  Self-reported average sitting hours per day: participants report number of hours (to the nearest whole hour) spent sitting on a typical workday.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Will adhere to data sharing regulations of target journal
Supporting Information: Study Protocol, SAP
Time Frame: Study registered online at clinical trials.gov (permanent). This includes statistical analysis plan. Data accessible on request - available for 7 years.
Access Criteria: Data accessible on request - available for 7 years.

REFERENCES:
- [Result] Blake H, Lai B, Coman E, Houdmont J, Griffiths A. Move-It: A Cluster-Randomised Digital Worksite Exercise Intervention in China: Outcome and Process Evaluation. Int J Environ Res Public Health. 2019 Sep 17;16(18):3451. doi: 10.3390/ijerph16183451. PMID 31533292